CLINICAL TRIAL: NCT06872619
Title: A Registry for Prostate Cancers
Brief Title: RegisterPROS - a Registry for Prostate Cancers
Acronym: RegisterPROS
Status: Enrolling by invitation | Type: Observational
Sponsor: Wren Laboratories LLC (Industry)
Collaborators: Münster University Hospital, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: WREN_REGISTER_02
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer (Adenocarcinoma); Prostate Biopsy; Prostatectomy; Radioligand; Chemotherapy; Androgen Deprivation Therapy; PSA
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection (RNA stabilization tube) used for prostate cancer biomarker measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prostate cancer subjects: Subjects at risk or who have a histological confirmation of prostate cancer disease (all Gleason grades, all stages including castration resistant disease). Interventions include ADT, chemotherapy and RLT
  Interventions: Device: PROSTest

INTERVENTIONS:
Device: PROSTest — Multianalyte Algorithm Analysis of circulating prostate cancer transcripts

SUMMARY:
Prostate cancers are derived from epithelial cells in the prostate gland. Treatment options include surgery, medical (androgen signaling targeted and chemotherapy) and radiation therapy including radioligand therapy (RLT). Survival is linked to early and accurate diagnoses or to the effective detection of disease recurrence and/or treatment failure. One challenge is to develop accurate non-invasive tests that can detect prostate cancer disease activity. A second challenge is to evaluate the effectiveness of such biomarkers during the natural history of this disease (e.g., active surveillance). A third aim is to identify whether molecular markers can predict response to different therapies (either pre-treatment, or early on during the first few cycles of a therapy). RegisterPROS registry aims at collecting data and blood samples from patients being evaluated for PCa disease. Data will be entered prospectively and anonymized after informed consent. All physicians who treat PCas are invited to participate to the registry. Data will be evaluated within regular time frames, focusing on diagnostic accuracy for biomarkers in the different types of tumors, treatment modalities and patient outcomes (e.g. disease recurrence and survival), thereby contributing to an understanding of the role of biomarkers in tumor management.

DETAILED DESCRIPTION:
Background: Survival of PCas is linked to early and accurate diagnoses of aggressive disease (GG2-5) and effective detection of disease progression and/or recurrence (minimal residual disease or treatment failure). Tissue based molecular markers have been developed and have utility (e.g., OncoType Dx). Blood-based markers e.g., ARV-7 detection may also have utility. However, PSA (and changes in levels from baseline) are considered the current standard of care. Molecular markers e.g., PROSTest, have been developed but little is known about the utility of these markers in clinical practice. Objective: To systematically and prospectively collect clinical information and samples (blood and saliva) from PCas in Europe, Africa, Caribbean and the USA based a histologically confirmed diagnosis. Methods: PCas will be enrolled and followed up following informed consent. Data will be entered prospectively and anonymized. Patient history are completed by contributing physicians and samples are collected for analysis. All information will be transferred to a database. Evaluation of treatment modalities and patient outcomes (e.g. disease recurrence) will be assessed at follow-up times. The primary objectives of the project are to:

1a) assess diagnostic accuracy of molecular-based blood tests e.g., PROSTest.

1. b) evaluate utility of molecular-based tests e.g., PROSTest to monitor PCa patients (active surveillance or on treatment).

   The secondary objectives of the project include:
2. a) assess utility of molecular-based tools to detect disease recurrence

2b) examine whether these tools can predict response to different therapies

Analyses will include:

1. Descriptive statistical analyses including demographics, histology and grading, treatment types.
2. Clinical follow-up and blood chemistry (PSA) and molecular results.
3. Correlation analyses between blood results and clinical data. This will include assessment of the time at which the results significantly (and consistently) increases and the time of tumor recurrence and an evaluation whether the change in blood results is predictive of disease recurrence and/or treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* All subjects

Exclusion Criteria:

* Female

Ages: 45 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a histologically confirmed diagnosis of a prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
PCa diagnosis | 5 years
  Histology confirmed prostate cancer disease
Surveillance | 10 years
  Natural progression of disease

SECONDARY OUTCOMES:
Minimal residual disease | 10 years
  Detection of MRD
Therapy efficacy | 10 years
  Treatment response assessment

CONTACTS AND LOCATIONS:
Overall Officials: Abdel Halim, PhD, PharmD, Study Director — Wren Laboratories; Kambiz Rahbar, MD, Principal Investigator — Munster University Hospital
Locations (1):
- University Hospital Munster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Modlin IM, Kidd M, Drozdov IA, Boegemann M, Bodei L, Kunikowska J, Malczewska A, Bernemann C, Koduru SV, Rahbar K. Development of a multigenomic liquid biopsy (PROSTest) for prostate cancer in whole blood. Prostate. 2024 Jun;84(9):850-865. doi: 10.1002/pros.24704. Epub 2024 Apr 3. PMID 38571290
- [Background] Rosin RD, Haynes A, Kidd M, Drozdov I, Modlin I, Halim A. Evaluation of a multigenomic liquid biopsy (PROSTest) for prostate cancer detection and follow-up in a Caribbean population. Cancer Epidemiol. 2024 Oct;92:102642. doi: 10.1016/j.canep.2024.102642. Epub 2024 Aug 9. PMID 39121520
- [Background] Rahbar K, Kidd M, Prasad V, David Rosin R, Drozdov I, Halim A. Clinical Sensitivity and Specificity of the PROSTest in an American Cohort. Prostate. 2025 May;85(6):558-566. doi: 10.1002/pros.24858. Epub 2025 Jan 21. PMID 39838708